CLINICAL TRIAL: NCT01318629
Title: Invasive Findings in Patients With Angina Equivalent Symptoms But No Coronary Artery Disease; Results From the Heart Quest Cohort Study
Brief Title: Angina in Non Coronary Artery Disease
Acronym: HeartQuest
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Prof. Paul Erne, Prof. Paul Erne, Luzerner Kantonsspital
Other Study IDs: Heart Quest
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Angina Pectoris; Microvascular Angina; Angina Pectoris, Variant
MeSH Terms: conditions — Angina Pectoris; Microvascular Angina; Angina Pectoris, Variant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many patients undergoing coronary angiography are found to have no significant coronary artery disease (CAD) despite angina equivalent symptoms and/or electrocardiographic abnormalities suggestive of myocardial ischemia. The aim of this study is to systematically assess patients with angina equivalent symptoms despite normal coronary angiograms and to evaluate their symptoms according to a defined algorithm.

DETAILED DESCRIPTION:
All consecutive patients who had coronary angiography at the Luzerner Kantonsspital between July 1st 1996 and July 31st 2008 and who had no significant coronary stenoses (no coronary stenoses ≥ 50%) were recruited for this study. Patients are extensively examined during angiography using acetylcholine infusion and fast atrial pacing. According to the result of the additional invasive examination (vasospasm, vasoconstriction, vasodilation; symptoms during examination) a distinct diagnosis is attributed to the patients (small vessel disease, vasospastic disease, hypertensive heart disease, rhythm disorder, or extracardiac thoracic pain including pulmonary hypertension). Patients are followed-up after 10 years and prognosis of these patients is assessed (including mortality, cardiovascular events, re-angiography, functional status after 10 years).

ELIGIBILITY:
Inclusion Criteria:

* Coronary angiography at the Luzerner Kantonsspital between July 1st 1996 and July 31st 2008
* No significant coronary stenoses (no coronary stenoses ≥ 50%)

Exclusion Criteria:

* Severe valvular heart disease
* Severe congestive heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who had coronary angiography at the Luzerner Kantonsspital between July 1st 1996 and July 31st 2008 and who had no significant coronary stenoses (no coronary stenoses ≥ 50%) were recruited for this study.
Sampling Method: Probability Sample
Enrollment: 718 (Actual)
Dates: Start 1996-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Cause of angina equivalent symptoms in patients with no coronary artery disease | One day
Prognosis of patients with angina equivalent symptoms and normal coronary arteries | 10 years after baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Schoenenberger AW, Adler E, Gujer S, Jamshidi P, Kobza R, Stuck AE, Resink TJ, Erne P. Prognostic value of an abnormal response to acetylcholine in patients with angina and non-obstructive coronary artery disease: Long-term follow-up of the Heart Quest cohort. Int J Cardiol. 2016 Oct 15;221:539-45. doi: 10.1016/j.ijcard.2016.07.035. Epub 2016 Jul 6. PMID 27414736
- [Derived] Schoenenberger AW, Felber S, Gujer S, Moser A, Jamshidi P, Stuck AE, Erne P. Invasive findings in patients with angina equivalent symptoms but no coronary artery disease; results from the heart quest cohort study. Int J Cardiol. 2013 Jul 15;167(1):168-73. doi: 10.1016/j.ijcard.2011.12.053. Epub 2012 Jan 10. PMID 22236508